CLINICAL TRIAL: NCT02895945
Title: A Phase 3, Multicenter, Open-label Study of the Efficacy and Safety of B-Domain Deleted Recombinant Porcine Factor VIII (BAX 802) in Subjects With Congenital Hemophilia A With Factor VIII Inhibitors Undergoing Surgical or Other Invasive Procedures
Brief Title: BAX 802 in CHA With Inhibitors
Acronym: CHAWI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Takeda has determined that the benefit/risk profile does not support continuation of the surgery Study for this specific Congenital Hemophilia A with Inhibitors patient population.
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 241502; 2015-005521-39 (EudraCT Number)
Record Dates: First submitted 2016-08-15; First posted 2016-09-12 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAX 802 in Surgery (Experimental): Participants who are undergoing major or minor elective surgical, dental, or other invasive procedures.
  Interventions: Biological: Antihemophilic Factor (Recombinant), Porcine Sequence (BAX 802)

INTERVENTIONS:
Biological: Antihemophilic Factor (Recombinant), Porcine Sequence (BAX 802) — In case of major surgery, FVIII target level is ≥80% for major surgeries/ procedures and ≥50% for minor surgeries/ procedures.
  Other Names: BAX 802; recombinant porcine factor VIII; Obizur; rpFVIII

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BAX 802 in males with congenital hemophilia A (CHA) with inhibitors who are undergoing major or minor elective surgical, dental, or other invasive procedures.

ELIGIBILITY:
Inclusion Criteria

1. Participant requires a major or minor elective surgical, dental or other invasive procedure
2. Participant is male and ≥ 12 to ≤ 75 years old at the time of screening
3. Participant has provided signed informed consent (and assent for adolescent participants, as applicable) in accordance with local regulatory requirements
4. Participant has severe (factor VIII (FVIII) level < 1%) or moderately severe (FVIII level ≤ 2%) congenital hemophilia A (CHA) with inhibitors to human factor VIII (hFVIII) of ≥ 0.6 Bethesda units (BU), as tested at screening at the central laboratory
5. Participant is not currently receiving or has recently received (< 30 days) immune tolerance induction (ITI) therapy
6. Participant has a Karnofsky performance score of ≥ 60 at screening
7. Participant is human immunodeficiency virus negative (HIV-); or HIV+ with stable disease and CD4+ count ≥ 200 cells/mm^3 at screening
8. Participant is hepatitis C virus negative (HCV-) by antibody or polymerase chain reaction (PCR) testing; or HCV+ with chronic stable hepatitis disease. Positive serologies will be confirmed by PCR testing.
9. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria

1. The participant requires emergency surgery
2. Severe chronic liver dysfunction or disease (e.g., ≥ 5 × upper limit of normal [ULN] alanine aminotransferase [ALT], as confirmed by central laboratory at screening or a documented prothrombin time/international normalized ratio [PT/INR] > 1.5)
3. Clinically symptomatic renal disease (serum creatinine > 2.0 mg/dL), as confirmed by central laboratory at screening
4. Anti-porcine factor VIII (pFVIII) inhibitor > 10 BU prior to surgery
5. Platelet count < 100,000/μL at screening
6. Participant has another active coagulation disorder, other than hemophilia A, as per the medical history
7. Planned use of α-interferon with or without ribavirin for HCV infected patients or planned use of a protease inhibitor for HIV infected patients. Patients currently taking any of these medications for ≥ 30 days are eligible
8. Known hypersensitivity to recombinant porcine factor VIII (rpFVIII), or hamster or murine proteins
9. Participant has an ongoing or recent (within 3 months of screening) thrombo-embolic disease, fibrinolysis or disseminated intravascular coagulation (DIC)
10. Participant has been exposed to an IP within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational product (IP) or investigational device during the course of this study
11. Participant is unable to tolerate quantity of blood to be drawn for protocol procedures
12. Participant is a family member or employee of the Investigator.

Ages: 12 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (23):
- United States (3):
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
- Bulgaria (2):
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - UMHATEM 'N.I. Pirogov', EAD, Sofia
- Hopital Maisonneuve-Rosemont d/b/a CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec, Canada
- Germany (2):
  - Universitaetsklinikum Bonn AoeR, Bonn
  - Zentrum für Hämostaseologie, Universitätsklinikum Leipzig AöR, Leipzig
- Italy (4):
  - Presidio Ospedaliero di Castelfranco Veneto, Castelfranco Veneto, Treviso
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Padova, Padua
- UMC Utrecht, Utrecht, Netherlands
- Oslo Universitetssykehus - Rikshospitalet, Oslo, Norway
- Instytut Hematologii i Transfuzjologii-1-1Y7-1347, Warsaw, Poland
- FSBI of Science "Kirov Scientific and Research Institute of Hematology and Blood Transfusion of FMBA., Kirov, Russia
- Bleeding Disorders Unit and Clinical Haematology Service at Charlotte Maxeke JHB Academic Hospital, Johannesburg, South Africa
- Spain (3):
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario La Paz, Madrid
- Turkey (Türkiye) (3):
  - Ankara University Medical Faculty, Ankara
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc64db2bf003ab45d54

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 sites in Italy, Netherlands, Poland, Germany and Turkey. Study was initiated on 22 December 2016 and terminated on 22 January 2021.
Pre-assignment Details: A total of 8 participants planned for Major Surgeries and Minor Surgeries received recombinant porcine factor VIII (rpFVIII) (BAX 802).
Groups:
- Major Surgeries: Male participants with congenital hemophilia A (CHA) with inhibitors to human factor VIII (hFVIII) undergone major surgical invasive procedures initially received loading dose BAX 802 infusion, intravenously to maintain a minimum target factor VIII (FVIII) level of greater than or equal to (>=) 80 percent (%) approximately 1 to 2 hours prior to the surgery. Subsequent dosing was based on participant's FVIII activity levels, body weight and investigator's clinical judgement.
- Minor Surgeries: Male participants with CHA with inhibitors to hFVIII undergone minor surgical invasive procedures initially received loading dose BAX 802 infusion, intravenously to maintain a minimum target FVIII level of >=50% approximately 1 to 2 hours prior to the surgery. Subsequent dosing was based on participant's FVIII activity levels, body weight and investigator's clinical judgement.
Period: Overall Study
Arm/Group | Major Surgeries | Minor Surgeries
Started | 7 | 1
SAS (Safety analysis set (SAS) comprised of all participants who received any amount of BAX 802.) | 7 | 1
FAS (Full analysis set (FAS) comprised of all participants with at least one available hemostatic assessment.) | 7 | 0
Completed | 5 | 0
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: SAS comprised of all participants who received any amount of BAX 802.
Groups:
- Major Surgeries: Male participants with CHA with inhibitors to hFVIII undergone major surgical invasive procedures initially received loading dose BAX 802 infusion, intravenously to maintain a minimum target FVIII level of >=80% approximately 1 to 2 hours prior to the surgery. Subsequent dosing was based on participant's FVIII activity levels, body weight and investigator's clinical judgement.
- Total: Total of all reporting groups
Arm/Group | Major Surgeries | Minor Surgeries | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (14.39) | 58.0 | 38.6 (15.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Surgeries With a "Good" or "Excellent" Response as Measured by the Global Hemostatic Efficacy Assessment (GHEA) Score
Description: GHEA score consisted of 3 individual rating scales: (1) Intra-operative Efficacy Assessment Scale, (2) Post-operative Efficacy Assessment Scale, and (3) Overall Peri-operative Efficacy Assessment Scale. Scales 1 and 2 was performed by the operating surgeon on Day 1, and Scale 3 was performed by the investigator on Day 14. Each rating scale was based on 4 points scale ranging from: 3 (Excellent), 2 (Good), 1 (Fair), and 0 (None). Total score ranged from 0 to 9, where scores evaluated as: excellent (7 to 9), good (5 to 7), fair (3 to 4), and none (0 to 2). The scores of 3 individual ratings scales were added together to form a GHEA score. For a GHEA score of 7 to be rated "excellent" with no individual assessment scores less than (<) 2 and at least 1 assessment score equal to (=) 3; otherwise a score of 7 was rated "good". Percentage of Surgeries With a "Good" or "Excellent" response as measured by the GHEA score were reported.
Time Frame: Day 1 up to discharge or Day 14 (whichever was earlier)
Population: Full analysis set (FAS) comprised of all participants with at least one available hemostatic assessment.
Measure: Number; unit: percentage of surgeries
Units Other Than Participants: surgeries
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 0
Number analyzed (surgeries) | 7 | 0
percentage of surgeries
  GHEA rating: Good | 14.3 |
  GHEA rating: Excellent | 71.4 |

2. Secondary Outcome: Actual Blood Loss, Estimated Volume of Expected Average Blood Loss and Expected Maximum Blood Loss During Intra-operative, Post-operative and Peri-operative Period
Description: Prior to the surgery, the surgeon/investigator predicted and compared the estimated volume (in milliliter [mL]) of the expected average blood loss and expected maximum blood loss for the planned surgical intervention in a comparable healthy individual with similar demographic characteristics; for intraoperative, postoperative, and overall perioperative time periods. Intra-operative defined as period from start of surgery to completion of surgical procedure. Post-operative defined as period from completion of surgical procedure till 24 hours post-surgery. Peri-operative defined as period from start of surgical procedure till discharge or 14 days post surgery (whichever was earlier). Actual blood loss, estimated volume of expected average blood loss and expected maximum blood loss during each operative period was reported.
Time Frame: Intra-operative: up to completion of surgery (Day 1), Post-operative: at 24 hours post-surgery, and Peri-operative: at discharge or Day 14 (whichever was earlier)
Population: FAS comprised of all participants with at least one available hemostatic assessment. Here "number analyzed" were participants who were evaluable for the outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Units Other Than Participants: surgeries
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 0
Number analyzed (surgeries) | 7 | 0
milliliter (mL)
  Intra-operative Period: Actual Blood Loss | 141.1 (188.69) |
  Intra-operative Period: Expected Average Blood Loss | 221.7 (286.76) |
  Intra-operative Period: Expected Maximum Blood Loss | 414.7 (546.37) |
  Post-operative Period: Actual Blood Loss: number analyzed (Participants) | 5 | 0
  Post-operative Period: Actual Blood Loss | 31.0 (66.56) |
  Post-operative Period: Expected Average Blood Loss | 171.4 (276.17) |
  Post-operative Period: Expected Maximum Blood Loss | 378.0 (570.94) |
  Peri-operative Period: Actual Blood Loss | 164.1 (215.15) |
  Peri-operative Period: Expected Average Blood Loss | 465.0 (744.85) |
  Peri-operative Period: Expected Maximum Blood Loss | 842.9 (1310.01) |

3. Secondary Outcome: Ratio of Actual Blood Loss and Estimated Volume of Expected Average Blood Loss During Intra-operative, Post-operative and Peri-operative Period
Description: Prior to the surgery, the surgeon/investigator predicted and compared the estimated volume (mL) of the expected average blood loss and expected maximum blood loss for the planned surgical intervention in a comparable healthy individual with similar demographic characteristics; for intraoperative, postoperative, and overall perioperative time periods. Intra-operative defined as period from start of surgery to completion of surgical procedure. Post-operative defined as period from completion of surgical procedure till 24 hours post-surgery. Peri-operative defined as period from start of surgical procedure till discharge or 14 days post surgery (whichever was earlier). Ratio of actual blood loss and estimated volume of expected average blood loss during each operative period was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: surgeries
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 0
Number analyzed (surgeries) | 7 | 0
ratio
  Intra-operative Period | 0.970 (0.9486) |
  Post-operative Period: number analyzed (Participants) | 5 | 0
  Post-operative Period | 0.150 (0.2236) |
  Peri-operative Period | 0.545 (0.3448) |

4. Secondary Outcome: Ratio of Actual Blood Loss and Expected Maximum Blood Loss During Intra-operative, Post-operative and Peri-operative Period
Description: Prior to the surgery, the surgeon/investigator predicted and compared the estimated volume (mL) of the expected average blood loss and expected maximum blood loss for the planned surgical intervention in a comparable healthy individual with similar demographic characteristics; for intraoperative, postoperative, and overall perioperative time periods. Intra-operative defined as period from start of surgery to completion of surgical procedure. Post-operative defined as period from completion of surgical procedure till 24 hours post-surgery. Peri-operative defined as period from start of surgical procedure till discharge or 14 days post surgery (whichever was earlier). Ratio of actual blood loss and expected maximum blood loss during each operative period was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: surgeries
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 0
Number analyzed (surgeries) | 7 | 0
ratio
  Intra-operative Period | 0.555 (0.6517) |
  Post-operative Period: number analyzed (Participants) | 5 | 0
  Post-operative Period | 0.058 (0.0846) |
  Peri-operative Period | 0.306 (0.1962) |

5. Secondary Outcome: Percentage of Major Surgeries With Good or Excellent Hemostatic Score
Description: Percentage of major surgeries with good or excellent hemostatic score was analyzed by GHEA score. It consisted of 3 individual ratings: (1) Intra-operative Efficacy Assessment Scale, (2) Post-operative Efficacy Assessment Scale, (3) Postoperative Efficacy Assessment Scale. Ratings 1 and 2 was performed by the operating surgeon on Day 1, and Rating 3 was performed by the investigator on Day 14. Each rating scale was based on 4 point scale ranging from: 3 (Excellent), 2 (Good), 1 (Fair), and 0 (None). The scores of each of the 3 individual ratings scales, was added together to form a GHEA score. Total score ranged from 0 to 9 where scores evaluated as excellent (7 to 9), good (5 to 7), fair (3 to 4), and none (0 to 2). Hemostatic efficacy success was defined as "excellent" or "good "outcome for >=70% of hemostatic efficacy assessments. Percentage of major surgeries with good or excellent hemostatic score were reported.
Time Frame: Day 1 up to discharge or Day 14 (whichever was earlier)
Population: FAS comprised of all participants with at least one available hemostatic assessment. As planned, this outcome measure was only analyzed for major surgeries. There were 7 participants analyzed for major surgeries and all the 7 participants underwent 7 surgeries.
Measure: Number (95% Confidence Interval); unit: percentage of surgeries
Units Other Than Participants: surgeries
Arm/Group | Major Surgeries
Number analyzed (Participants) | 7
Number analyzed (surgeries) | 7
percentage of surgeries | 85.7 [42.1 to 99.6]

6. Secondary Outcome: Average Daily Weight-adjusted Dose of BAX 802 Per Participant During Pre-operative, Intra-operative and Post-operative Period
Description: Body-weight adjusted dose equals to amount infused/body-weight (kilogram [kg]), where amount infused as amount of drug infused (International Units [IU]) and body-weight as the last available body-weight (kg) prior to the infusion. Pre-operative defined as period prior to surgery. Intra-operative defined as period from start of surgery to completion of surgical procedure. Post-operative defined as period from completion of surgical procedure till discharge or 14 days post surgery (whichever was earlier). Average daily weight-adjusted dose of BAX 802 per participant during each operative period was reported.
Time Frame: Pre-operative: before surgery, Intra-operative: up to completion of surgery (Day 1), Post-operative: from completion of surgical procedure till discharge or 14 days post surgery (whichever was earlier)
Population: SAS comprised of all participants who received any amount of BAX 802. Here "number analyzed" were participants who were evaluable for the outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: International Units per kilogram (IU/kg)
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
International Units per kilogram (IU/kg)
  Pre-operative | 162.471 (125.7051) | 208.779
  Intra-operative: number analyzed (Participants) | 6 | 0
  Intra-operative | 76.083 (35.1339) |
  Post-operative: number analyzed (Participants) | 7 | 0
  Post-operative | 43.549 (56.0039) |

7. Secondary Outcome: Total Weight-adjusted Dose of BAX 802 Per Participant During Pre-operative, Intra-operative and Post-operative Period
Description: Body-weight adjusted dose equals to amount infused/body-weight (kg), where amount infused as amount of drug infused (IU) and body-weight as the last available body-weight (kg) prior to the infusion. Pre-operative defined as period prior to surgery. Intra-operative defined as period from start of surgery to completion of surgical procedure. Post-operative defined as period from completion of surgical procedure till discharge or 14 days post surgery (whichever was earlier). Total weight-adjusted dose of BAX 802 per participant during each operative period was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
IU/kg
  Pre-operative | 162.471 (125.7051) | 208.779
  Intra-operative: number analyzed (Participants) | 6 | 0
  Intra-operative | 76.083 (35.1339) |
  Post-operative: number analyzed (Participants) | 7 | 0
  Post-operative | 625.520 (399.4913) |

8. Secondary Outcome: Volume of Blood Products Transfused
Description: The volume (in mL) of blood products transfused from initiation of the intervention to discharge or Day 14 (whichever came earlier) was reported.
Time Frame: From initiation of the surgery up to discharge or Day 14 (whichever came earlier)
Population: FAS comprised of all participants with at least one available hemostatic assessment. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 2 | 0
mL | 950.0 (70.71) |

9. Secondary Outcome: Number of Participants With De Novo Inhibitors
Description: De novo inhibitor was defined as a post-baseline inhibitor titer to FVIII (hFVIII or porcine factor VIII [pFVIII])of >=0.6 Bethesda units per milliliter (BU/mL) given a baseline of <0.6 BU/mL. Number of participants with de novo inhibitors were reported.
Time Frame: Baseline up end of study (EOS) (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants
  hFVIII | 0 | 0
  pFVIII | 3 | 0

10. Secondary Outcome: Number of Participants With Anamnestic Reactions
Description: An anamnestic reaction was defined as an increase from a measurable baseline (>0.6 BU/mL) in the inhibitor titer to FVIII (human or porcine) of >=10 BU/mL. Number of participants with anamnestic reactions were reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants
  hFVIII | 5 | 0
  pFVIII | 3 | 0

11. Secondary Outcome: Mean Change From Baseline up to EOS in Inhibitory and Binding Antibodies to pFVIII
Description: The assessment of inhibitory antibodies (immunoglobulin G [IgG] and immunoglobulin M [IgM]) to pFVIII was determined using Bethesda assay, and assessment of binding antibodies (IgG and IgM) to pFVIII was determined using validated enzyme-linked immunosorbent assays (ELISAs). Mean change from baseline in inhibitory and binding antibodies to pFVIII was reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: BU/mL
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 6 | 1
BU/mL | 111.15 (149.072) | -0.20

12. Secondary Outcome: Mean Change From Baseline up to EOS in Inhibitory and Binding Antibodies to hFVIII
Description: The assessment of inhibitory antibodies (IgG and IgM) to hFVIII was determined using Bethesda assay, and assessment of binding antibodies (IgG and IgM) to hFVIII was determined using ELISA. Mean change from baseline in inhibitory and binding antibodies to hFVIII was reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: BU/mL
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 6 | 1
BU/mL | 198.67 (317.254) | -0.20

13. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Binding Antibodies to Baby Hamster Kidney (BHK) Proteins
Description: The assessment of binding antibodies to BHK proteins was determined using ELISA. Clinical significance was judged by the investigator. Number of participants with clinically significant change from baseline in binding antibodies to BHK proteins were reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Thromboembolic Events
Description: Thromboembolism defined as formation in a blood vessel of a clot (thrombus) that breaks loose and carried by the blood stream to plug another vessel. Number of participants with thromboembolic events was reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Severe Allergic Reactions
Description: Number of participants with severe allergic reaction (example: anaphylaxis) after administration of study drug were reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Investigational Product (IP) Related Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Serious AE was any untoward medical occurrence (whether considered to be related to study assigned treatment or not) that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in a congenital abnormality/birth defect, or was an important medical event. TEAEs was defined as any adverse events (classified by preferred term) that had a start date on or after the first dose of study treatment or that had a start date before the date of first dose of study treatment, but increased in severity after the first dose of study treatment. TEAEs included both serious and non-serious TEAEs.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants
  IP related TEAEs | 4 | 0
  IP related serious TEAEs | 4 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign
Description: Vital sign parameters included: temperature, pulse rate, respiration rate, systolic and diastolic blood pressure. Any changes in vital signs which were deemed clinically significant was judged by the investigator. Number of participants with clinically significant change from baseline in vital signs were reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Values
Description: Clinical laboratory assessment included hematology and clinical chemistry. Any changes in clinical laboratory results which were deemed clinically significant was judged by the investigator. Number of participants with clinical significant change from baseline in clinical laboratory values were reported.
Time Frame: Baseline up to EOS (up to 44 months)
Population: SAS comprised of all participants who received any amount of BAX 802.
Measure: Count of Participants; unit: Participants
Arm/Group | Major Surgeries | Minor Surgeries
Number analyzed (Participants) | 7 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to EOS (up to 44 months)
Arm/Group | Major Surgeries | Minor Surgeries
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/7 | 0/1
Other Adverse Events (participants affected / at risk) | 3/7 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Surgeries (N=7) | Minor Surgeries (N=1)
Anamnestic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Anti factor VIII antibody increased (Investigations) | 2 (2) | 0 (0)
Anti factor VIII antibody positive (Investigations) | 3 (3) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Surgeries (N=7) | Minor Surgeries (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was discontinued as Takeda determined that the benefit/risk profile did not support continuation of the surgery study for this specific Congenital Hemophilia A with Inhibitors participant population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT02895945/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT02895945/SAP_001.pdf